CLINICAL TRIAL: NCT00511485
Title: Protocol EC-FV-03: A Phase II Study of EC145 in Patients With Progressive Adenocarcinoma of the Lung
Brief Title: Study of Vintafolide (MK-8109, EC145) in Participants With Progressive Adenocarcinoma of the Lung (MK-8109-008, EC-FV-03)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8109-008; EC-FV-03 (Other: Endocyte)
Record Dates: First submitted 2007-08-02; First posted 2007-08-06 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Adenocarcinoma of the Lung
Keywords: Cancer; Adenocarcinoma; Phase II; Lung; Non-small cell lung cancer; NSCLC; EC145; EC20
MeSH Terms: conditions — Adenocarcinoma of Lung; Neoplasms; Adenocarcinoma; Carcinoma, Non-Small-Cell Lung | interventions — EC145; technetium 99m etarfolatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Etarfolatide + Vintafolide (Experimental): Screening: After completion of all screening procedures and confirmation of eligibility, all participants receive a 1- to 2-mL injection of 0.1 mg etarfolatide labeled with 20 to 25 mCi of technetium-99m. Induction phase of treatment: Two 4-week cycles; if stable disease or better at (week 8) computed tomography (CT), participant may proceed into maintenance phase. Maintenance phase of treatment: 4-week cycles with CT every 8 weeks. Participants continue on study until they experience disease progression, unacceptable toxicity, or attain protocol-defined clinical benefit.
  Interventions: Drug: Vintafolide; Drug: Etarfolatide

INTERVENTIONS:
Drug: Vintafolide — Induction: vintafolide 1.0 mg intravenous injection, Monday through Friday, for the first 3 weeks of each 4 week cycle. Maintenance: vintafolide 2.5 mg intravenous injection, Monday, Wednesday, and Friday, weeks 1 and 3 of each 4 week cycle. At the investigator's discretion, participants may receive vintafolide via an ambulatory pump after the first week of therapy has been administered in the clinic setting.
Drug: Etarfolatide

SUMMARY:
This is a Phase II clinical trial evaluating the benefit from therapy with vintafolide in participants with progressive adenocarcinoma of the lung.

DETAILED DESCRIPTION:
This is a Phase II clinical trial of vintafolide administered to participants with progressive adenocarcinoma of the lung.

Vintafolide is a drug that is specifically designed to enter cancer cells via the folate vitamin receptor (FR). Experimental evidence shows that this target receptor is expressed on a significant portion of non-small cell lung cancers. Early clinical evidence in a small number of Phase I patients suggests that vintafolide is generally well-tolerated, without many of the side-effects observed in more-standard therapeutic agents. This evidence suggests that vintafolide may be useful as a chemotherapy against progressive adenocarcinomas of the lung. The primary objective of this study is to collect data on clinical benefit produced by therapy with vintafolide .

All participants will undergo imaging with the FR targeting investigational imaging agent etarfolatide (EC20, FolateScan) during the screening period to confirm eligibility for the treatment portion of the clinical trial. Clinical evidence suggests that etarfolatide may be used to identify patients with cancers that express the target receptor.

Information about the safety and tolerability of both vintafolide and etarfolatide will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, progressive, adenocarcinoma of the lung.
* Previously received at least 2 cytotoxic containing chemotherapeutic regimens (can include an epidermal growth factor receptor [EGFR] inhibitor). There is no upper limit to the number of prior chemotherapeutic regimens.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* At least 4 weeks from prior therapy and recovered from associated acute toxicities.
* Radiographic evidence of measurable disease and ertafolide "positive" tumor.
* Adequate bone marrow reserve, hepatic, and renal function.
* Negative serum pregnancy test for women of childbearing potential and willingness to practice contraceptive methods.

Exclusion Criteria:

* Serious comorbidities (as determined by the Principal Investigator).
* History of carcinomatous peritonitis.
* History of severe bowel obstruction (as determined by the Principal Investigator).
* Women who are pregnant or lactating.
* Prior radiation therapy to assessable disease, unless disease progression is confirmed at that site.
* Participants requiring palliative radiotherapy at time of study entry.

Note: Participants with central nervous system (CNS) metastasis are eligible if a) they have been treated for the CNS metastasis and have been clinically stable (with regard to their CNS disease) for >4 weeks and b) they do not require steroids or antiseizure medications (i.e., for seizure control), or if the CNS metastasis has been untreated to date, it is not associated with a midline shift or significant edema and there is no clinically-evident requirement for steroids or antiseizure medication. In either situation, participants must be off steroids and/or antiseizure medications for at least 14 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Percentage of patients deriving clinical benefit | Clinical benefit is defined as the ability to receive 4 or more cycles (i.e., months) of therapy without progression of disease.

SECONDARY OUTCOMES:
Tumor responses to EC145 therapy | Duration of EC145 therapy will vary according to individual participant response.
Progression-free survival, response duration, and overall survival time observed after EC145 therapy | 2 years after completing therapy with EC145 and the 30-day follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Binh Nguyen, MD, PhD, Study Director — Endocyte

REFERENCES:
- [Background] Reddy JA, Dorton R, Westrick E, Dawson A, Smith T, Xu LC, Vetzel M, Kleindl P, Vlahov IR, Leamon CP. Preclinical evaluation of EC145, a folate-vinca alkaloid conjugate. Cancer Res. 2007 May 1;67(9):4434-42. doi: 10.1158/0008-5472.CAN-07-0033. PMID 17483358